CLINICAL TRIAL: NCT02900963
Title: Nutritional Assessment of Locally Advanced Head and Neck Cancer Patients Who Underwent Exclusive or Adjuvant Radiotherapy or Chemo-radiotherapy
Brief Title: Nutritional Status Assessment in Head and Neck Cancer Patients Receiving Radiotherapy or Chemo-radiotherapy
Acronym: NUTRINECK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB 13.04
Record Dates: First submitted 2016-07-28; First posted 2016-09-15 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Head and Neck Cancer
Keywords: Nutrition; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutrition state determination (Other): Determination of nutritional state and inflammatory status:
  weekly assessment of patient's weight biological parameters (albumin, transthyretin, orosomucoid) and weekly assessment of patient's weight
  Interventions: Other: weekly assessment of patient's weight

INTERVENTIONS:
Other: weekly assessment of patient's weight — Biological assessment to determine biological and inflammatory status Quality of life questionary

SUMMARY:
Radiotherapy and chemotherapy are standard treatment of head and neck cancer alone or associated to surgical treatment. Early (during treatment or the following weeks) and late side effects contribute to malnutrition in this population at risk. In this context, nutritional support adapted by dietary monitoring and enteral nutrition (nasogastric tube or gastrostomy) are often necessary. The early identification of the patients with high malnutrition risk and requiring enteral nutrition is necessary to improve the tolerance and efficacy of treatment. This prospective study research the factors of malnutrition during head and neck radiotherapy.

DETAILED DESCRIPTION:
Head and neck cancer is one of the most common malignancies in the world, Malnutrition occurs frequently at the time of diagnosis as consequences of alcohol consumption and tobacco use that is quite common in this patients population, and of local tumor invasion, obstructing the function of swallowing and chewing. In addition, during the treatment, mucositis, anorexia, dysphagia, mouth sores, and other acute and late toxic effects of radiotherapy (RT) and chemotherapy frequently worsen the nutritional status.

Poor nutritional status and chemotherapy or RT-toxicity, lead to treatment interruption frequently and is also associated with higher risk of infection, hospital readmission, early death, worse survival outcomes, and deterioration in the quality of life (QoL). According to published results, one third of the patient would have benefit from a complete treatment. In addition, the correlation exists between some biological parameters (CRP, albumin, neutrophils, Hb) and the nutritional status. Therefore, it deems essential to maintain nutritional status in head and neck cancer patients undergoing RT and chemotherapy.

Dietary counseling and oral supplements showed positive influences on nutritional outcomes and QoL However, their role is limited when it comes to obstruction or mucositis. Thus, enteral feeding may be a choice either through nasogastric tube (NGT) or percutaneous endoscopic gastrostomy (PEG). Studies investigated the effects of PEG compared with NGT were not conclusive or showing no consistent results on nutritional status, treatment interruption, nutrition-related hospital admission, and tube-related complications in the head and neck cancer patients receiving RT or chemo-radiotherapy.

The optimal method and the timing of placement are still debated. Consequently, the aim of this study is to collect data on our current daily practice on supplementary nutrition method ( NGT, PEG) in head and neck cancers patients treated in our radiation therapy unit and to identify factors predicting good treatment outcomes( ie full treatment administration).

Secondary objectives are to collect nutritional data during the treatment, to study the nutritional status in relation to acute or late adverse events, to study the impact of an early enteral feeding on clinical and biological parameters.

Ancillary study: Sarco-Nutrineck The aim of this ancillary study is to collect data on prevalence of low muscle mass in this population, treatment outcomes and survival.

Study measures:

At baseline: body height and weight, calculated BMI. Biological parameters: albumin, orosomucoid, transthyretin, CRP Daily - during the treatment period: weight Weekly - during the treatment period: albumin, orosomucoid, transthyretin, CRP. The Nutritional and inflammatory status score will be calculated.

Clinical criteria on the requirement of enteral nutrition (or need for artificial nutrition) in case of weight loss persisting at least for three days during radiotherapy:

The aim of this study is to investigate whether nutritional screening on admission can be used to determine risk levels for adverse clinical events and treatment outcome ( full treatment administration) in head and neck cancer and to propose a risk stratification based on nutritional screening before radiotherapy or concomitant chemo radiotherapy.

tube (NGT) will be placed according to the following procedure: The weight will be assessed on daily basis and will be compared to the figure at baseline, before treatment. If the weight loss is superior to 2 kg, the patient will consult a radiotherapist who will perform a physical examination, a nutritional assessment (history, appetite change, taste, quantity and quality of oral food intake, medication, details regarding weight change and BMI). In addition to dietary counselling and oral supplementation, If indicated, analgesic drugs and or treatment of associated mucositis will be prescribed.

In case of persisting weight loss or severe dysphagia or no oral solid food intake, a nasogastric tube (NGT) will be placed by a nurse and a personalized nutritional counselling by a dietician will be organized.

Biological exams will be done according to our local practice and standard, and the results will be analyzed to assess the safety. Regular clinical exams will be realized. All adverse events will reported according to the common terminology criteria for adverse events scale.

Follow-up period. The patients will benefit from a clinical exam, height, weight, BMI, biological exam (including albumin, orosomucoid, transthyretin, CRP) one month after the end of the treatment, and then at three months and at twelve months, late toxicities will be recorded.

The aim of this study is to investigate whether nutritional screening on admission can be used to determine risk levels for adverse clinical events and treatment outcome (full treatment administration) in head and neck cancer and to propose i) isk stratification based on nutritional screening before radiotherapy or concomitant chemo radiotherapy ii) decisional algorithm on placement of a NGT

ELIGIBILITY:
Inclusion Criteria:

* Males or females older than 18 years
* Performance Status 0 or 1 or 2
* Locally advanced head and neck cancer treated with a curative intent treatment consisting of either concomitant chemo-radiotherapy or adjuvant radiation therapy or adjuvant chemo-radiotherapy.
* Signed Informed Consent

Exclusion Criteria:

* Other cancer or previous cancer within 2 years or evolutive cancer
* Performance Status 3 or 4
* NGT or PEG at screening period
* Any legal, social, psychological reasons that could jeopardize the patient's compliance to the study constrains.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2014-04; Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
weight | one year
  Measure of weight ( in Kg)

SECONDARY OUTCOMES:
Nutritional status determination | 3 months
  Determination of nutritional status by assessing albuminemia
Nutritional status determination | 3 months
  Determination of nutritional status by assessing transthyretin
Nutritional status determination | 6 months
  Determination of nutritional status by assessing albuminemia
Nutritional status determination | 6 months
  Determination of nutritional status by assessing transthyretin
Nutritional status determination | One year
  Determination of nutritional status by assessing albuminemia
Nutritional status determination | One year
  Determination of nutritional status by assessing transthyretin
Inflammatory status | 3 months
  Determination of inflammatory status by assessing orosomucoid
Inflammatory status | 3 months
  Determination of inflammatory status by assessing CRP
Inflammatory status | 6 months
  Determination of inflammatory status by assessing orosomucoid
Inflammatory status | 6 months
  Determination of inflammatory status by assessing CRP
Inflammatory status | one year
  Determination of inflammatory status by assessing orosomucoid
Inflammatory status | one year
  Determination of inflammatory status by assessing CRP
BMI calculation | one year
  Calculation of BMI using height and weight

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Thureau, MD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No